CLINICAL TRIAL: NCT00769665
Title: A 2-week Clinical Comparison of SYSTANE® Ultra to Sensitive Eyes Rewetting Drops in Contact Lens Wearing Patients.
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: SMA-08-15
Record Dates: First submitted 2008-10-07; First posted 2008-10-09 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Dry Eye; re-wetting drops
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Systane Ultra: Systane Ultra
  Interventions: Other: Systane Ultra
- Sensitive Eyes: Sensitive Eyes
  Interventions: Other: Sensitive Eyes Rewetting Drops

INTERVENTIONS:
Other: Systane Ultra — Re-wetting ocular eye drop
  Groups: Systane Ultra
Other: Sensitive Eyes Rewetting Drops — Re-wetting ocular eye drop
  Groups: Sensitive Eyes

SUMMARY:
To evaluate safety with the use of Systane Ultra in contact lens wearers. A comparison to a currently marketed contact lens rewetting drop will be included as a control.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 18 and 65 years of age.
* Provide written Informed Consent.
* Must be wearing a planned replacement soft lens in a 2 week or monthly replacement modality, or a Rigid Gas Permeable (RGP) contact Lens
* Must have best corrected distance visual acuity, with contact lenses, of 20/30 or better in each eye.
* Sodium fluorescein (NaFl) corneal staining score sum of < 2 in both eyes (NEI scoring system).
* Must be willing to maintain pre-enrollment systemic medication regimens during the study.
* Must be available for study visits and to fill out study questionnaires.

Exclusion Criteria:

* Has modified their systemic medications within 30 days prior to enrollment.
* Has a history of allergy to any study product ingredients
* Is unwilling or unable to meet the study visit timeline.
* Has any active corneal, eyelid or other anterior segment inflammation or infection, which, in the opinion of the Investigator, would adversely affect successful contact lens wear.
* Is currently using any topical eye medications (not including rewetting drops, artificial tear products or Restasis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2008-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events and Visual Acuity | 2 weeks